CLINICAL TRIAL: NCT05779982
Title: Outcomes of Sentinel Node Biopsy According to MRI Response in an Association With the Subtypes in cN1-3 Breast Cancer After Neoadjuvant Systemic Therapy
Brief Title: SURPASS Retrospective Study
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Gwe Ahn, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2022-0362
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Breast MRI; Neoadjuvant Systemic Therapy; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multicenter retrospective cohort: This study included patients diagnosed with breast cancer who received neoadjuvant systemic therapy (NAST) followed by curative surgery between January 2013 and December 2018. All patients were cN1-3 breast cancer at initial presentation confirmed by any imaging studies (either ultrasonography or MRI) or pathological examination using ultrasonography-guided needle biopsy of suspicious axillary lymph nodes. The clinical nodal stage was determined based on findings from physical examination, with imaging studies such as ultrasonography or MRI taken into account, according to the American Join Committee on Cancer guidelines (7th edition). In addition, all patients underwent sentinely lymph node biopsy (SLNB) followed by axillary lymph node dissection. SLNB was performed using a radioactive marker, blue dye, or both (dual tracers).
  Interventions: Procedure: Sentinel lymph node biopsy followed by axillary lymph node dissection

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy followed by axillary lymph node dissection — This is a retrospective study to determine the feasibility of sentinel lymph node biopsy (SLNB) after neoadjuvant systemic therapy (NAST) according to response to NAST and breast cancer subtypes. All patients received SLNB followed by axillary lymph node dissection after NAST.

SUMMARY:
This study aimed to determine whether sentinel lymph node biopsy (SLNB) could be a reliable option for evaluating nodal status in patients who had responded well to neoadjuvant systemic therapy (NAST), even if they had initially presented with a high nodal burden. The study investigated the outcomes of SLNB followed by axillary lymph node dissection (ALND) in this patient population, taking into account the response to NAST and the breast cancer subtype.

DETAILED DESCRIPTION:
To determine the feasibility of sentinel lymph node biopsy (SLNB) in this study, the investigators evaluated the false-negative rate (FNR) of SLNB. The FNR was calculated as the number of patients with negative SLNs who had a residual disease in the rest of the axillary lymph nodes (ALNs) divided by the total number of patients with residual disease in either the SLNs, the rest of the ALNs, or both: FN/true-positive + FN. The investigators compared the FNR of the SLNB according to the radiologic response measured using breast MRI in each subtype. The investigators further evaluated the FNR in subgroups stratified by clinical nodal stage. Additionally, the investigators assessed additional metastatic ALNs in cases with 1-2 metastatic SLNs through the completion of ALN dissection.

ELIGIBILITY:
Inclusion Criteria:

* cN1-3 breast cancer at initial presentation
* received neoadjuvant systemic therapy (NAST)
* received sentinel lymph node biopsy (SLNB) followed by additional axillary lymph node dissection (ALND)
* breast MRI performed at baseline and post-NAST.

Exclusion Criteria:

* case with unavailable data for breast MRI and operation

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients diagnosed with breast cancer who received neoadjuvant systemic therapy (NAST) followed by curative surgery between January 2013 and December 2018. All patients were cN1-3 breast cancer at initial presentation In addition, all patients underwent sentinely lymph node biopsy (SLNB) followed by axillary lymph node dissection.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
False negative rate of sentinel lymph node biopsy according to radiologic response stratified by brest cancer subtype | up to 1 month after the breast surgery
  False negative rate of sentinel lymph node biopsy according to radiologic response stratified by brest cancer subtype

SECONDARY OUTCOMES:
False negative rate of sentinel lymph node biopsy according to clinical nodal stage | up to 1 month after the breast surgery
  False negative rate of sentinel lymph node biopsy according to clinical nodal stage
Additional axillary lymph node metastasis rate in patients with 1-2 metastatic sentinel lymph nodes | up to 1 month after the breast surgery
  Additional axillary lymph node metastasis rate in patients with 1-2 metastatic sentinel lymph nodes

IPD SHARING:
Plan to Share IPD: Undecided